CLINICAL TRIAL: NCT00300937
Title: Coenzyme Q10 Supplementation in Pregnant Women as Strategy to Reduce Maternal Morbidity Due to Preeclampsia
Brief Title: Coenzyme Q10 Supplementation and Development of Preeclampsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teran, Enrique, MD, PhD (Individual)
Collaborators: Ecuadorian Foundation for Science and Technology - FUNDACYT (Unknown); Universidad Central del Ecuador (Other); Jarrow Formulas Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PFN-03-053
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — 100 mg oral BID starting at week 20 until delivery

SUMMARY:
As preeclampsia is a disease specially affecting young and primiparous women, and due to the fact that we found previously in several studies a prevalence of 12%, to ensure a confidence of 95% and a power of 80%, it is necessary to include a total of 190 women (95 in each arm), therefore it is planned to recluse a total of 200 pregnant women currently attending to the outpatients clinic at the HGOIA for pregnancy control before than week 20 of gestation.

From each one of those women the clinical research team will obtain an obstetric, anthropometric and clinical record following the current regulations of the Ecuadorian Public Health Ministry. All women included will be under a detailed prenatal control every 4 weeks from week 20 of pregnancy, this will include gestational age, weight, umbilical perimeter, uterine altitude, fetal cardiac frequency and maternal blood pressure.

In addition, in each schedule visit an urine test will be done (to discard proteinuria), also a venous blood sample (10 ml) in heparinized tubes will be taken and immediately transported to the Biomedical Center for centrifugation and plasma isolation. During week 20, all women will be assigned (using a randomized numbers table) to one of the following groups: a) intervention group, that will received two capsules of 100 mg of coenzyme Q10 twice daily up to delivery; or b) control group, that will receive two capsules of the correspondent placebo twice daily up to delivery. Both, active and placebo capsules will be manufactured by the same provider (Jarrow Formulas, Los Angeles, CA, USA) to guarantee that weight, size, odor and color are similar.

Absolutely all women participating in the study will know all contact information of the clinical team and will be allowed to request medical care as frequent as they needed, independently of establish obstetrical controls. Preeclampsia diagnosis will be performed only by clinical researchers and based on a persistent high blood pressure higher than 140/90 mmHg and proteinuria higher than 300 mg/24 hours.

Coenzyme Q10 will be measured using a high performance liquid chromatography equipment (HPLC) and the method previously described and validated by our group.

The hypothesis is that in the group receiving CoQ10 supplementation will be less cases of preeclampsia compared to placebo.

DETAILED DESCRIPTION:
This research will be conducted in collaboration between the Experimental Pharmacology and Cellular Metabolism at the Biomedical Center in the Central University of Ecuador and the Department of Obstetric Pathology in the Gynecology and Obstetrics Hospital "Isidro Ayora" (HGOIA) in Quito, Ecuador. It is proposed a descriptive, prospective, double blind, randomized and placebo controlled experimental study to identify cause-effect rather than effectiveness of the treatment in which, after approval of the Bioethics Committee (COBI) of the Biomedical Center as well as the Bioethics Committee of the HGOIA, each one of the possible women to be included in the study, after a careful and detailed lecture and explanation about the objectives and procedures by one of the researchers will be invited to take a part in it and will be asked to sing the respective inform consent.

As preeclampsia is a disease specially affecting young and primiparous women, and due to the fact that we found previously in several studies a prevalence of 12%, to ensure a confidence of 95% and a power of 80%, it is necessary to include a total of 190 women (95 in each arm), therefore it is planned to recluse a total of 200 pregnant women, primigravidae, younger than 25 years old and with no history of diseases related to the cardiovascular, endocrine, metabolic nor reproductive systems, who were currently attending to the outpatients clinic at the HGOIA for pregnancy control before than week 20 of gestation. Those women with positive inclusion criteria and who accepted to participate in the study will be randomized to one of the treatment groups.

From each one of those women the clinical research team will obtain an obstetric, anthropometric and clinical record following the current regulations of the Ecuadorian Public Health Ministry. Women with history of hypertension, currently taken any kind of medication, or that not want to participate in the study will be excluded. All women included will be under a detailed prenatal control every 4 weeks from week 20 of pregnancy, this will include gestational age, weight, umbilical perimeter, uterine altitude, fetal cardiac frequency and maternal blood pressure. These information will be collected into the clinical record of the HGOIA and in a special designated form useful for later data entry in an electronic database (Epi Info V6.04).

In addition, in each schedule visit an urine test will be done (to discard proteinuria), also a venous blood sample (10 ml) in heparinized tubes will be taken and immediately transported to the Biomedical Center for centrifugation and plasma isolation. Plasma aliquots of 500 ul will be frozen at -80°C up to the analysis. During all this process samples will be protected from direct light with aluminum foil and from extreme temperatures with a refrigerated flask. Samples received at the Biomedical Center will be identified only with a code; therefore biochemical analysis will be also performed in a blind fashion. During week 20, all women will be assigned (using a randomized numbers table) to one of the following groups: a) intervention group, that will received two capsules of 100 mg of coenzyme Q10 twice daily up to delivery; or b) control group, that will receive two capsules of the correspondent placebo twice daily up to delivery. Both, active and placebo capsules will be manufactured by the same provider (Jarrow Formulas, Los Angeles, CA, USA) to guarantee that weight, size, odor and color are similar. The different bottles for those women will be prepared by a member of the team not related to the clinical control of women, and a careful control of the number of tablets in each bottle will be taken to later on analyze the accomplishment of the treatments. The blind codes will be obtained before the intervention started and will be responsibility of the principal investigator up to the end of the study.

Absolutely all women participating in the study will know all contact information of the clinical team and will be allowed to request medical care as frequent as they needed, independently of establish obstetrical controls. In addition, as a part of the study their attention in the HGOIA will be mandatory. Preeclampsia diagnosis will be performed only by clinical researchers and based on a persistent high blood pressure higher than 140/90 mmHg measured two times with the patient rested for at least 10 minutes and with a mercury sphygmomanometer two times (Riester, Germany) and proteinuria higher than 300 mg/24 hours or two crosses in a diskstip with 3-24 hours apart.

Coenzyme Q10 and alpha tocopherol will be measured using a high performance liquid chromatography equipment (HPLC) and the method previously described and validated by our group. In brief, plasma samples will be processed in an HPLC equipped with a reverse phase ODS-C18 column (5 um, 150x4.6 mm) with its respective guard column (5 um, 10x4.6 mm). Mobile phase will be methanol/ethanol (40:60 v/v) previously filtered and with a continuous flow of 1ml/min. The UV detector will be set up to a wavelength of 275 nm. Samples (0.5 ml) will be mixed with 0.5 ml of sodium dodecyl sulphate (SDS) at 20% and 50 ul of CoQ9 solution in ethanol as internal standard. Later will be added 2 ml of a methanol/propanol solution (95:5 v/v) and will be vorterex vigorously by 30 seconds, after that, 5 ml of hexane will be added and vorterex again by 60 seconds. Organic and aqueous solvents will be separated by centrifugation at low speed (1000 g by 5 min). Four and half ml of the organic phase will be transferred to another vial and dissecatted under continuous nitrogen flow and then reconstituted with ethanol. Prepared samples will be immediately analyzed and kept all the time under ice and protected form light. Measurements will be performed in duplicate and average values will be used for the statistical analysis. Intra and inter assay variation coefficients, as well as recover percentage will be calculate to ensure the uniformity of the assays. Also, total cholesterol, as well as, low and high cholesterol lipoproteins will be measured using a spectrophotometer.

Primary endpoint will be the number of preeclampsia cases in each group, and the severity of the disease and quality of the newborn (weight, height, cephalic perimeter and gestational age at born).

ELIGIBILITY:
Inclusion Criteria:

* Primigravidae
* Younger than 25 years old
* No history of disease related to cardiovascular, endocrine, metabolic or reproductive systems
* To be recruited before than week 20 of gestation
* To sign the Informed Consent form

Exclusion Criteria:

* Voluntary withdrawal
* Poor compliance of visit/treatment

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 235 (Actual)
Dates: Start 2004-07; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Preeclampsia rate in both groups | Delivery

SECONDARY OUTCOMES:
Newborns weight | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Teran, MD, PhD, Study Director — Biomedical Center - Central University of Ecuador
Locations (1):
- Hospital Gineco-obstetrico Isidro Ayora, Quito, Ecuador